CLINICAL TRIAL: NCT06337695
Title: VERIFY: Vedolizumab for the Prevention of Immune Checkpoint Inhibitor Related Diarrhea or Colitis in Patients With Cancer: A Randomized, Double-Blinded, Placebo Controlled Trial
Brief Title: VERIFY: Vedolizumab for the Prevention of Immune Checkpoint Inhibitor Related Diarrhea or Colitis in Patients With Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HREBA.CC-23-0271
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Cancer Metastatic
Keywords: Immune Checkpoint Inhibitors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — vedolizumab

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blinded, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vedolizumab (Experimental): Participants receive 300 mg vedolizumab IV at weeks 0, 3, 6, 14, and 22.
  Interventions: Biological: Vedolizumab
- Placebo (Placebo Comparator): Participants receive 300 mg placebo IV at weeks 0, 3, 6, 14, and 22.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Vedolizumab — 300 mg IV at weeks 0, 3, 6, 14, and 22
  Arms: Vedolizumab
Biological: Placebo — 300 mg IV at weeks 0, 3, 6, 14, and 22
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the prevention of immune checkpoint inhibitors (ICIs) related diarrhea/colitis using vedolizumab in participants with unresectable stage III or metastatic stage IV cancer, starting standard of care (SOC) immunotherapy

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo up to a 2-week screening period to confirm their eligibility. Eligible patients will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Vedolizumab or placebo and given their first dose within 2 weeks of starting their SOC immunotherapy. Vedolizumab or placebo will be administered at Weeks 0, 2, 6, 14, and 22.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study specific activities or procedures
* Diagnosed with unresectable advanced stage III or metastatic stage IV malignancy
* Planned for initiation of SOC immunotherapy and development of prognostic biomarker evidence that predisposes to ICI diarrhea/colitis risk
* Ability to and willingness to adhere to the randomized treatment interventions (vedolizumab or placebo), administered intravenously

Exclusion Criteria:

* Condition(s) for which vedolizumab is contraindicated (e.g., hypersensitivity reaction, known allergic reaction to vedolizumab or its components)
* Current or prior use of vedolizumab or prior immunotherapy exposure for cancer
* Presence of inflammatory bowel disease (Crohn's disease, ulcerative colitis), indeterminate colitis, or microscopic colitis
* Presence of ileostomy, colostomy, or short bowel syndrome
* Presence of known luminal gastrointestinal metastases at baseline
* Presence of significant pre-existing autoimmune disease (at investigator's discretion)
* Presence of severe infection(s) or opportunistic infection(s)
* Active enteric infection with viral, bacterial, or parasitic pathogens
* Presence of untreated latent or active tuberculosis, or untreated chronic hepatitis B virus
* Baseline ECOG status grade ≥3
* Pregnancy or lactation
* Treatment with another investigational product within 8 weeks of randomization
* Requirement for baseline anti-diarrheal treatment(s) (including but not limited to loperamide, diphenoxylate-atropine, octreotide, tincture of opium), anticholinergic drug(s), or opioid-based analgesic(s) used specifically for diarrhea control within 14 days of randomization
* Any condition or diagnosis, that could in the opinion of the Qualified Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hazard Ratio of Patients achieving ICI-related diarrhea and colitis-free survival a 6-months | Start of immunotherapy therapy and for 6 months
  ICI-related diarrhea and colitis will be assessed using Common Terminology Criteria for Adverse Events (CTCAE), and a grade ≥2 will be considered an event.

SECONDARY OUTCOMES:
Proportion of patients with histologically confirmed colitis-free survival at 6 months | 6 months
  Colitis-free survival will be defined as CTCAE grade ≥2 based on a biopsy taken at time of patient meeting the primary endpoint or at 6 months.
Proportion of patients with severe diarrhea or colitis at 6 months | 6 months
  Severe diarrhea or colitis will be defined as CTCAE grade ≥3
Hazard Ratio of patients with diarrhea or colitis after 6 months | 6-12 months
  Diarrhea or colitis will be defined as CTCAE grade ≥2
Total average dose of checkpoint inhibitor therapy received within 6 and 12 months | 0 to 6 months; and 0 to 12 months
  The total average dose of ICI therapy will be used
Proportion of participants who require temporary ICI discontinuation due to immune-related adverse events (irAEs) | 0 to 12 months
  Temporary discontinuation of ICI therapy will be defined as any delay of 1-week or more resulting from an immune-related adverse event (irAE), as identified and graded using the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Proportion of participants who require permanent ICI discontinuation due to irAEs | 0 to 12 months
  Permanent discontinuation of ICI therapy will be defined as stopping ICI therapy, and not restarting within the 1-year time window of the trial resulting from an immune-related adverse event (irAE), as identified and graded using the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Proportion of patients requiring rescue corticosteroids for ICI related diarrhea/colitis | at 6-months and 12-months
  Any patient who receives rescue corticosteroids within the first 6 months or within the first 12 months will be considered an event.
Total average prednisone equivalent dose of rescue corticosteroids required | at 6-months and 12-months
  The prednisone equivalent dose will be calculated using the following conversions:
  Cortisone 5mg = Prednisone 1mg Hydrocortisone 4mg = Prednisone 1mg Prednisolone 1mg = Prednisone 1mg Methylprednisolone 0.8mg = Prednisone 1mg Dexamethasone 0.15mg = Prednisone 1mg
Proportion of participants requiring all-cause hospitalization by Day +180 and Day +365 | at day 180 and 365
  Chart review will be used to identify hospitalizations.
Proportion of participants requiring ICI-related diarrhea/colitis-specific hospitalization by Day +180 and Day +365 | at day 180; at day 365
  Chart review will be used to identify hospitalization and determine the cause of hospitalization.
Mean change in the EuroQol EQ-5D instrument at Day +180 and Day +365 compared to baseline | baseline to day 180; baseline to day 365
  The EuroQol EQ-5D is a validated questionnaire for patients with inflammatory bowel disease.
Overall survival (measured as death) at +180 and Day +365 compared to baseline | Day +180 and Day +365
  All-cause mortality will be used to compare the survival rate of the therapy and placebo arms. The rates will be calculated for 6 months (defined at day 180) and 1-year (day 365).
Progression-free survival at 6- and 12-months, defined using the Response Evaluation Criteria in Solid Tumors (RECIST), v1.176 | At Day +180 and Day +365
  Progression-free survival will be defined using the Response Evaluation Criteria in Solid Tumors (RECIST), v1.176
Proportion of participants experiencing any adverse events (AEs) | At Day +180 and Day +365
  Adverse events will be defined as described in good clinical practice.
Proportion of participants experiencing serious AEs | At Day +180 and Day +365
  Serious adverse events will be defined as described in good clinical practice.
Proportion of participants experiencing other irAEs | At Day +180 and Day +365
  Adverse events will be defined as described in good clinical practice. Those that are immune related will be used for this outcome.